CLINICAL TRIAL: NCT01055275
Title: Cook Iliac Branch Graft Post-market Registry
Status: Terminated | Type: Observational
Why Stopped: Terminated due to low enrollment.
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-016
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Iliac Aneurysm; Aortic Aneurysm
Keywords: iliac aneurysm; aortic aneurysm; endovascular grafts
MeSH Terms: conditions — Iliac Aneurysm; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cook Iliac Branch Graft: Patients implanted with a Cook Iliac Branch Graft
  Interventions: Device: Implantation with a Cook Iliac Branch Graft

INTERVENTIONS:
Device: Implantation with a Cook Iliac Branch Graft — Treatment of an aortic, aorto-iliac or iliac aneurysm with a CE-marked Cook Iliac Branch Graft.

SUMMARY:
The Cook Iliac Branch Graft Post-market Registry will obtain case reports of physician experience with a CE-marked Cook Iliac Branch Graft to further confirm device safety and performance.

ELIGIBILITY:
Inclusion Criteria:

* CE-Marked Cook Iliac Branch Graft (e.g., Zenith® Branch Endovascular Graft-Iliac Bifurcation, Zenith® Helical Branch Endovascular Graft)
* Registry data are de-identified with respect to patient.

Exclusion Criteria:

* Patient for whom this device would not normally be considered standard of care.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with a Cook Iliac Branch Graft.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Internal iliac artery patency | 1 year
Aneurysm Exclusion | 1 year

SECONDARY OUTCOMES:
Death | 1 year
Conversion | 1 year
Rupture | 1 year
Success Measures | 1 year
Major Complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Riambau, MD, PhD, Principal Investigator — Hospital Clinic, Barcelona, Spain
Locations (1):
- Hospital Clinic, Barcelona, Spain